CLINICAL TRIAL: NCT05516134
Title: All About Me: An Intervention to Ease the Transition to Long-term Care, Build Community, and Improve Quality of Care for Persons With Dementia
Brief Title: All About Me: An Intervention to Ease the Transition to Long Term Care
Acronym: AAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopeful Aging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG077993-01
Record Dates: First submitted 2022-08-10; First posted 2022-08-25 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Dementia; Alzheimer Disease; Dementia, Vascular; Dementia, Mixed; Dementia of Alzheimer Type
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Mixed Dementias

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants who receive the intervention (all)
  Interventions: Behavioral: SAFE at Home

INTERVENTIONS:
Behavioral: SAFE at Home — The All About Me (AAM) app will consist of Serious Digital Health Games for PWD. The market-ready version of the app will consist of five components. (1) The Fun Facts About Me Game will be used when a PWD is moving into LTC. The goal of the game is to provide an enjoyable way for family members and PWD to provide important information about the PWD's background. (2) The Resident Game Bundle will consist of SDHGs that will allow PWD to learn about one another in an enjoyable way. (3) The My Residents Module will provide staff with a convenient way to view information about a PWD with whom they will be working. Staff will launch this module from any device. (4) The Meet the Staff Module, which will be developed and tested in a future Phase II study, will allow residents to learn about staff members at their community. (5) The AAM Training Modules will provide staff and family members with access to video-based training modules that describe how to use relevant portions of the app

SUMMARY:
This Phase I study will involve initial development and evaluation of an innovative cross-platform software app called All About Me (AAM), which will consist of Serious Digital Health Games (SDHGs) for PWD. The AAM app will assist staff in providing person-centered care and enable residents to improve relationships with one another and with staff, thereby promoting a sense of community. This Phase I study has three Specific Aims: (1) Develop an Alpha version of the AAM App, (2) Examine acceptability of and satisfaction with the AAM App, and (3) Examine the impact of the Resident Game Bundle / Survey Says Game on engagement/affect.

DETAILED DESCRIPTION:
Study Design: The study will utilize a quasi-experimental pre-post design.

Sample:

PWD: Twenty-four PWD will take part in the study, including 12 ALF residents and 12 living in a NH.

Family Members: Twenty-four family members will also take part in the study-i.e., one for each PWD. In some cases, the "family member" may be a friend or legally authorized representative.

Staff Members: Twelve LTC staff members will take part in the quasi-experiment-five at the ALF and five at the NH.

Inclusion/Exclusion Criteria:

PWD must reside in an ALF or NH, be 60+ years old, speak and read English, be diagnosed with dementia (of any type), and score at least eight on the MMSE.

Family Members, LTC Staff Members, and Focus Group Staff Members must be 18+ years old and speak and read English.

Baseline Period/Measures:

PWD: During Month 8, the following data will be collected via chart review: demographics, medications, diagnoses (including type of dementia), and primary language. In addition, the MMSE48 and the Dementia Quality of Life Scale (DEMQOL)50 will be administered via direct interview. The Neuropsychiatric Inventory-Nursing Home (NPI-NH),51,52 done via staff interview, will be used to collect data on challenging behaviors. PWD will also be observed taking part in standard activities using the Menorah Park Engagement Scale (MPES).53 The MPES is an observational scale that measures four types of engagement: Constructive Engagement (motor/verbal behavior exhibited clearly in response to the target activity); Passive Engagement (listening/watching a target activity); Distracted Engagement (motor/verbal behavior exhibited in response to something other than the target activity); and Non-Engagement/Apathy (outward signs/indicators of apathy, such as sleeping, closing one's eyes, and staring into space). The MPES also measures Pleasure, defined as clearly observable smiling/laughing. MPES data for standard activities will allow us to conduct a robust comparison to the RGB/Survey Says Game.

Family Members: researchers will interview family members to obtain demographics.

LTC Staff Members: Researchers will only interview staff members to obtain demographics during Phase I. Since this study is about development and feasibility testing, we do not want to unnecessarily burden staff with measures in Phase I. In the future Phase II, we will use the Caregiving Difficulty Scale-Intellectual Disability (CDS-ID)54 and the Maslach Burnout Inventory (MBI).

Intervention Period/Measures: During Month 9, family members will play the FFAM Game with their loved one on an Android tablet. A relatively lengthy four-week time period was chosen to ensure that even very busy family members will find time to play the game. We expect the game to take 60 minutes to complete, but we will encourage family members to split up the game into two 30-minute sessions. The app will automatically capture data about how many questions/items were completed and the length of time to complete the game. In addition, after playing the FFAM Game, family members and PWD will be asked questions related to ease of use and satisfaction. During Month 10, PWD will play the RGB/Survey Says Game twice per week for four weeks. The game will be played on an Android tablet, which will be connected to a large screen TV. The activity will be facilitated by a researcher; however, each staff member will observe an RGB/Survey Says Game session at least once, so that they can provide feedback about the game. An RA (not the researcher facilitating game) will observe PWD with the MPES while they are taking part in the Survey Says Game. After each Survey Says Game session, PWD and Staff Members will be asked questions related to ease of use and satisfaction (e.g., did you find the game easy to use? Did you enjoy the game? Would you recommend it to others?) During this same time period, LTC staff members will use the MRM daily when working with PWD. Each staff member will be given an Android smartphone and they will be encouraged to briefly review information about PWD before interacting with and/or providing care to them. At the end of this time period, staff will be asked questions related to ease of use and satisfaction for the MRM (e.g., Did you find it easy to use? Would you recommend it to others? Did it help you provide better care?)

Treatment Fidelity/Process Measures: In the backend of the app, a variety of treatment fidelity/process measures will automatically be collected by the app, including dates/times each participant used the app, length of time for each session; number of buttons pressed in each activity, and dates/times of any crashes.

Post-Treatment/Distal Measures:

PWD: The DEMQOL and NPI-NH will be re-administered. Family Members: No post-treatment measures will be taken. LTC Staff Members: No post-treatment measures will be taken.

Please note that, since the purpose of Phase I is to demonstrate proof of concept and feasibility, and since the intervention period will be relatively brief, changes are not expected from baseline to post-treatment on longer-term measures (i.e., the DEMQOL and NPI-NH). These measures are being used in Phase I exclusively to obtain means and standard deviations to conduct a power analysis to ensure that a sufficiently sized sample is used in Phase II.

Analyses: The AAM App will be considered successful if the following results are found: (1) at least 85% of participants complete 85% of the FFAM Game; (2) mean completion time for the FFAM Game is 45-75 minutes; (3) at least 85% of family members and PWD are satisfied with the FFAM Game and find it easy to use; (4) for PWD, levels of positive engagement/affect are higher, and levels of negative engagement are lower, during the Survey Says Game, as compared to standard programming (based upon a paired sample t-test); with the proposed sample size, and using means and standard deviations from the previous studies by the PI, we will have a power of 93% to detect effects (alpha = .05; one-tailed test). (5) at least 85% of PWD and LTC staff members are satisfied with the Survey Says Game and find it easy to use; and (6) at least 85% of LTC staff members are satisfied with the My Resident Module and find it easy to use.

ELIGIBILITY:
Inclusion Criteria:

* must be 60+ years old
* must speak and read English
* must have a clinical diagnosis of dementia (of any type)
* must score at least eight on the Mini-Mental Status Examination (MMSE)

Exclusion Criteria:

-shows signs of rapid physical / cognitive decline over the past six months, as indicated by medical records

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Skrajner, MA, Principal Investigator — Hopeful Aging
Locations (1):
- Hopeful Aging, Winchester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Participants with dementia who received the intervention. The intervention is called All About Me (AAM, which consists of Serious Digital Health Games for PWD, includuing the The Fun Facts About Me Game and the Resident Game Bundle (e.g., Survey Says).
- Family Members: These are family members who participated with their loved one in the study's intervention
- Staff Members: These are staff members who took the training and provided feedback about the training / intervention.
Period: Overall Study
Arm/Group | Treatment | Family Members | Staff Members
Started | 26 | 9 | 16
Completed | 25 | 9 | 16
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Persons With Dementia Who Recieved the Intervention: Participants who receive the intervention (all)
  SAFE at Home: The All About Me (AAM) app will consist of Serious Digital Health Games for PWD. The market-ready version of the app will consist of five components. (1) The Fun Facts About Me Game will be used when a PWD is moving into LTC. The goal of the game is to provide an enjoyable way for family members and PWD to provide important information about the PWD's background. (2) The Resident Game Bundle will consist of SDHGs that will allow PWD to learn about one another in an enjoyable way. (3) The My Residents Module will provide staff with a convenient way to view information about a PWD with whom they will be working. Staff will launch this module from any device. (4) The Meet the Staff Module, which will be developed and tested in a future Phase II study, will allow residents to learn about staff members at their community. (5) The AAM Training Modules will provide staff and family members with access to video-based training modules that describe how to use relevant portions of the app
- Family Members Who Participated in the Intervention With Their Loved One: This is a co-participant, family members who participated with their loved one in the study. Only some family members of participants were available to participate with their loved one. This is why there are more persons with dementia than family membeers
- Staff Members: These are staff members who took the training and gave feedback about the intervention
- Total: Total of all reporting groups
Arm/Group | Persons With Dementia Who Recieved the Intervention | Family Members Who Participated in the Intervention With Their Loved One | Staff Members | Total
Number analyzed (Participants) | 26 | 9 | 16 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.8 (10.2) | 68.9 (13.4) | 41.6 (14.1) | 68.5 (21.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 14 | 32
  Male | 14 | 3 | 2 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 26 | 9 | 15 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 0 | 8 | 17
  White | 15 | 9 | 8 | 32
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 9 | 16 | 51

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Treatment for Constructive Engagement on the Menorah Park Engagement Scale
Description: Constructive Engagement on the Menorah Park Engagement Scale is defined as doing or commenting on something related to the target activity. During baseline, multiple observations of "standard" activities were observed and a mean was calculated. Then, again, during treatment, multiple activities were observed and a mean was calculated. The minimum value for Constructive Engagement is zero (0) and the maximum score is two (2). Higher scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 21
score on a scale | 0.83 (0.45)
Statistical Analysis 1: Comparison: Treatment; baseline vs. treatment, paired sample t-test; Test type: Superiority; p < 0.01, t-test, 2 sided

2. Primary Outcome: Change From Baseline to Treatment for Passive Engagement on the Menorah Park Engagement Scale
Description: Passive Engagement on the Menorah Park Engagement Scale is defined as listening or watching something related to the target activity. During baseline, multiple observations of "standard" activities were observed and a mean was calculated. Then, again, during treatment, multiple activities were observed and a mean was calculated. The minimum value for Passive Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 21
score on a scale | 1.2 (0.86)
Statistical Analysis 1: Comparison: Treatment; Test type: Superiority; p < .01, t-test, 2 sided

3. Primary Outcome: Change From Baseline to Treatment for Other Engagement on the Menorah Park Engagement Scale
Description: Other Engagement on the Menorah Park Engagement Scale is defined as doing, commenting, listening, or watching something NOT related to the target activity. During baseline, multiple observations of "standard" activities were observed and a mean was calculated. Then, again, during treatment, multiple activities were observed and a mean was calculated. The minimum value for Other Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 21
score on a scale | -1.24 (0.78)
Statistical Analysis 1: Comparison: Treatment; Test type: Superiority; p < .01, t-test, 2 sided

4. Primary Outcome: Change From Baseline to Treatment for Non-Engagement on the Menorah Park Engagement Scale
Description: Non-Engagement on the Menorah Park Engagement Scale is defined as sleeping and/or staring into space. During baseline, multiple observations of "standard" activities were observed and a mean was calculated. Then, again, during treatment, multiple activities were observed and a mean was calculated. The minimum value for Non-Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 21
score on a scale | -.17 (0.34)
Statistical Analysis 1: Comparison: Treatment; Test type: Superiority; p = .03, t-test, 2 sided

5. Primary Outcome: Change From Baseline to Treatment for Pleasure on the Menorah Park Engagement Scale
Description: Pleasure on the Menorah Park Engagement Scale is defined as clearly observable laughing or smiling. During baseline, multiple observations of "standard" activities were observed and a mean was calculated. Then, again, during treatment, multiple activities were observed and a mean was calculated. The minimum value for Pleasure is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 21
score on a scale | .31 (.35)
Statistical Analysis 1: Comparison: Treatment; Test type: Superiority; p < .01, t-test, 2 sided

6. Secondary Outcome: Change From Baseline to Treatment on Dementia Related Quality of Life (DEMQOL)
Description: The Dementia Related Quality of Life Scale is a 28 item scale that examines quality of life in persons with dementia. The score ranges for 28 to 112. Higher scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Post-Treatment (Week 11)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 25
score on a scale | 2.40 (7.16)
Statistical Analysis 1: Comparison: Treatment; Test type: Superiority; p = .11, t-test, 2 sided

7. Secondary Outcome: Change From Baseline to Treatment on the Neuropsychiatric Inventory-Nursing Home (NPI-NH), Frequency x Severity Score (FxS)
Description: The NPI-NH examines 10 types of neuropsychiatric symptoms in persons with dementia, with the FxS score looking creating a composite score that takes into account frequency and severity of the symtoms. The score ranges from 0 to 120. Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Post-Treatment (Week 11)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 25
score on a scale | -9.1 (12.2)
Statistical Analysis 1: Comparison: Treatment; Test type: Superiority; p < .01, t-test, 2 sided

8. Secondary Outcome: Change From Baseline to Treatment on the Geriatric Depression Scale-Short Form (GDS-SF)
Description: The 15-item Geriatric Depression Scale (GDS-SF) is a screening tool used to assess depressive symptoms in older adults. Each item is answered with a "Yes" or "No"** response, with a total score ranging from 0 to 15, where higher scores indicate greater depressive symptoms. A score of 5 or more** suggests possible depression, warranting further clinical evaluation.
Time Frame: Baseline (Weeks 1-4) and Post-Treatment (Week 11)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 25
score on a scale | -0.97 (2.8)
Statistical Analysis 1: Comparison: Treatment; Test type: Superiority; p = 0.09, t-test, 2 sided

9. Secondary Outcome: Satisfaction With the App
Description: Satisfaction with the app
Time Frame: Treatment (Weeks 5-11)
Measure: Number; unit: % who said they were satisfied (yes/no)
Arm/Group | Treatment | Family Members | Staff Members
Number analyzed (Participants) | 26 | 9 | 16
% who said they were satisfied (yes/no) | 96 | 100 | 100

ADVERSE EVENTS:
Time Frame: 11 weeks
Description: Long-term care communities were asked to let the Principal Investigator (PI) know (via email, phone, or in person) about adverse events if/when they occur. In addition, each long-term care community was contacted via email at the end of each month by the PI. In that email, the PI asked the long-term care community whether any adverse events occurred that had not yet been reported. Staff and family members were also assessed for events, but not the target of the intervention.
Groups:
- Family Members: family members who played game with person with dementia
- Staff Members: staff who took training and gave feedback about the app
Arm/Group | Treatment | Family Members | Staff Members
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/9 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/9 | 0/16
Other Adverse Events (participants affected / at risk) | 0/26 | 0/9 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT05516134/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT05516134/SAP_001.pdf